CLINICAL TRIAL: NCT00574743
Title: A 12-month, Single-blind, Randomized, Parallel Group, Multicenter Study to Investigate the Efficacy and Safety of ERL080A Compared With MMF in de Novo Heart Recipients
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in Comparison to Mycophenolate Mofetil (MMF) in de Nove Heart Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CERL080A2401
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Heart Transplantation
Keywords: ERL080A, Heart Transplantation, Mycophenolate, EC-MPS

ARMS (2):
- 2 (No Intervention)
- 1 (Active Comparator)
  Interventions: Drug: Enteric-coated Mycophenolate Sodium

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate Sodium
  Arms: 1

SUMMARY:
This study will evaluate the safety and efficacy of EC-MPS (ERL080) in comparison to MMF in de novo heart recipients.

ELIGIBILITY:
Inclusion criteria

* Male or female cardiac patients 18-65 years old undergoing primary heart transplantation treated with CS-ME and corticosteroids as basic immunosuppression.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment. Effective contraception must be used during the trial and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility.
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion criteria

* Patients with donor hearts greater than 60 years of age and/or with cold ischemia time of more than 6 hours and/or donor hearts which have obvious coronary disease or are known to have heart disease at time of transplant.
* Patients on Left Ventricular Assist Device who have received any immunotherapy prior to transplantation or who are scheduled to receive immunotherapy thereafter.
* Patients with Panel Reactive Antibodies (PRA) 25%.
* Patients with serum creatinine 3.0mg/dL..
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.
* Patients with a history of significant coagulopathy or medical condition requiring long term anti-coagulation after transplantation (low aspirin treatment is allowed).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2002-01; Primary Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (9):
- United States (3):
  - Novartis Investigative site, Los Angeles, California
  - University of Minnesota, Minneapolis, Minnesota
  - Novartis Pharmaceuticals, Philadelphia, Pennsylvania
- Argentina (2):
  - Argentina, Buenos Aires
  - Site 1: X5000BJH, Córdoba
- Novartis Investigative site, Sydney, Australia, Sydney, Australia
- Canada (3):
  - Novartis Investigative, Edmonton, Alberta
  - Novartis, Toronto, Ontario
  - Novarits, Ottawa